CLINICAL TRIAL: NCT07316946
Title: Effects of Neuromuscular Taping on Shoulder Pain and Function in Pitchers: A Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sandra Jiménez-del-Barrio (Other)
Responsible Party: Sponsor-Investigator, Sandra Jiménez-del-Barrio, PhD Physiotherapist, University of Valladolid
Organization: University of Valladolid (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REF CEIm
Record Dates: First submitted 2025-12-09; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Pain
Keywords: neuromuscular taping; pain; function; shoulder
MeSH Terms: conditions — Shoulder Pain; Pain

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial 2 arms
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assessors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): The placebo group will receive the same bandage, with the same strip arrangement, but without any tension (0%) applied to any of the strips. Furthermore, participants will not receive any instructions for muscle activation during application. This placebo technique has been used in previous studies, supporting its methodological validity.
  Interventions: Other: Placebo Group
- Experimental group (Experimental): The experimental group will receive neuromuscular taping with kinesiology tape, consisting of two longitudinal strips applied along the lower trapezius muscle, with a tension close to 100% of the tape's elastic capacity. During application, the participant will be asked to activate the scapular depressor and retractor muscles.
  Additionally, two more longitudinal strips will be applied from the anterior portion of the humeral head towards the scapular spine, also with a tension close to 100%. During this application, the participant will be asked to activate the rotator cuff by applying a posteroanterior push to the humeral head.
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — The experimental group will receive a multilayer neuromuscular taping application using kinesiotape, consisting of the placement of two longitudinal strips in the direction of the lower trapezius, applied with tension close to 100% of the tape's elastic capacity. During the application, participants will be asked to activate the scapular depressor and retractor muscles.
  Additionally, two other longitudinal strips will be applied from the anterior portion of the humeral head toward the scapular spine, also with tension close to 100%. During this application, participants will be asked to activate the rotator cuff through a posteroanterior push of the humeral head.
  Arms: Experimental group
Other: Placebo Group — The placebo group will receive the same taping, with an identical arrangement of the strips, but without applying any tension (0%) to them. In addition, participants will not receive any instructions regarding muscle activation during the application. This placebo taping model has been used in previous studies, supporting its methodological validity.
  Arms: Placebo group

SUMMARY:
Effects of Neuromuscular Taping on Shoulder Pain and Function in Pitchers: A Clinical Trial

DETAILED DESCRIPTION:
Randomized clinical trial 2 arms

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* compete in a sport that involves overhead movement patterns
* train at least 2 hours per week
* shoulder pain lasting more than six weeks
* shoulder pain related to sports activity
* understand Spanish fluently enough to complete the questionnaire assessment.

Exclusion Criteria:

* presence of red flags that could suggest fractures, dislocations, or complete tendon ruptures, among others
* neurological pathologies
* other severe pathologies such as inflammatory arthritis, frozen shoulder
* having received corticosteroid injections or physiotherapy treatment in the last six months
* presence of previous surgeries
* pregnancy
* cognitive deficits that could limit the comprehension of the questionnaires or the physical evaluation
* skin problems that would be a contraindication for any type of bandage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-02-13 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Actual Pain Intensity | Baseline, after 30 minutes of the intervention and 72 hours after intervencion
  Pain intensity will be assessed using a 10-cm visual analog scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Participants will be asked to rate the intensity of pain experienced at the time of measurement
Pain Intensity during the arm elevation | Baseline, 30 minutes after intervention and 72 hours after intervention
  Pain intensity will be assessed using a 10-cm visual analog scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Participants will be asked to rate the intensity of pain experienced during arm elevation.

SECONDARY OUTCOMES:
Static Scapular Position | Baseline, 30 minutes after intervention and 72 hours after intervention
  Scapular position will be measured using an anterior/posterior scale. This static position will be recorded while standing, using a digital clinometer installed on a smartphone (Clinometer app). The inclinometer will be positioned directly over the scapular spine in the direction of the infraglenoid fossa.
Range of Motion | Baseline, 30 minutes after intervention and 72 hours after intervention
  Pain-free ROM during shoulder flexion, adduction, internal rotation, and external rotation will be measured following the protocol described by Shin et al.Participants will be instructed to flex the affected arm as far as possible, keeping the thumb pointing toward the ceiling. For adduction measurement, the patient will be placed in the side-lying position, and the evaluator will manually stabilize the scapula against the patient's thorax, allowing the arm to hang horizontally in adduction. For internal and external rotation, participants will be positioned supine with the shoulder abducted to 90°, the elbow flexed to 90°, and the forearm in a neutral position. A rolled towel will be placed under the humerus to maintain shoulder alignment. Participants will be asked to rotate their arm until pain onset or until scapular movement is observed. Three attempts of each movement will be recorded, and the mean range of motion (ROM) will be used for statistical analysis.
Functional Capacity | Baseline, 30 minutes after intervention and 72 hours after intervention
  Functional capacity will be assessed using the SPADI questionnaire. The SPADI is a patient-reported outcome measure designed to assess shoulder pain and functional disability. It consists of 13 items divided into two domains: pain and disability. The total score will be calculated by summing both domains and converting the result to a scale of 0 to 100, where higher scores indicate greater pain and disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Soria, Soria, Spain

IPD SHARING:
Plan to Share IPD: Undecided